CLINICAL TRIAL: NCT01933542
Title: The Effect of Chlorzoxazone on Moderate to Severe Postoperative Pain After Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Rikke Vibeke Nielsen, MD, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM2-RS-2013
Record Dates: First submitted 2013-08-23; First posted 2013-09-02 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Chlorzoxazone; Postoperative Pain
Keywords: Chlorzoxazone; Postoperative pain; Spine surgery; Opioid consumption
MeSH Terms: conditions — Pain, Postoperative | interventions — Chlorzoxazone; Morphine; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chlorzoxazone (Active Comparator): * Oral administration of chlorzoxazone 500 mg (two 250 mg tablets)
  * Morphine. Patient controlled intravenous morphine (PCA-pump), bolus 2.5 mg, lock-out-time 10 minutes. Concentration : Morphin 1 mg/ml.
  * Zofran 4 mg iv in case of moderate to severe nausea, supplemented by Zofran 1 mg iv if needed
  Interventions: Drug: Chlorzoxazone; Drug: Morphine; Drug: Zofran
- Placebo (Placebo Comparator): * Oral administration of two placebo tablets
  * Morphine. Patient controlled intravenous morphine (PCA-pump), bolus 2.5 mg, lock-out-time 10 minutes. Concentration : Morphin 1 mg/ml.
  * Zofran 4 mg iv in case of moderate to severe nausea, supplemented by Zofran 1 mg iv if needed
  Interventions: Drug: Placebo; Drug: Morphine; Drug: Zofran

INTERVENTIONS:
Drug: Placebo — Two placebo tablets identical to the chlorzoxazone tablets.
  Arms: Placebo
Drug: Chlorzoxazone — Two 250 mg chlorzoxazone tablets
  Arms: Chlorzoxazone
Drug: Morphine — Patient controlled intravenous morphine (PCA-pump), bolus 2.5 mg, lock-out-time 10 minutes. Concentration : Morphin 1 mg/ml.
Drug: Zofran — Zofran 4 mg iv. in case of moderate to severe nausea, supplemented by Zofran 1 mg iv. if needed

SUMMARY:
Chlorzoxazone is a centrally acting muscle relaxant used to treat muscle spasm and the resulting pain or discomfort. It acts on the spinal cord by depressing reflexes. Our purpose is to investigate the effect of chlorzoxazone on moderate to severe postoperative pain after spine surgery. Our hypothesis is that chlorzoxazone can reduce postoperative pain and reduce opioidconsumption and side effects compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing spine surgery in general anaesthesia.
* Postoperative pain > 50 mm on the VAS scale during mobilization.
* Patients who have not received analgesia 1 hour prior to inclusion.
* ASA 1-3.
* BMI > 18 og < 40.
* Fertile women need a negative HCG urine test.
* Patients who have given their written consent to participate and understand the contents of the protocol.

Exclusion Criteria:

* Participation in another clinical trial.
* Patients who do not speak and/or understand Danish.
* Fertile women with a positive HCG urine test.
* Allergy to the drugs used in the trial.
* Alcohol or medicine abuse, assessed by investigator.
* Daily use of strong opioids (morphine, ketobemidone, oxynorm, methadone, fentanyl)
* Daily chlorzoxazone treatment.
* Known or suspected porphyria.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Painscore during mobilization | 2 hours after taking the trial medication
  Painscore during active mobilization (VAS scale) defined by a standarized movement from recumbent position to sitting on the bedside

SECONDARY OUTCOMES:
Morphine consumption | 0-4 hours after taking the trial medication
  Total morphine consumption 0-4 hours after taking the trial medication, administered as patient controlled analgesia (PCA, bolus 2.5 mg, lockout 10 minutes).
Painscore during rest | 1, 2, 3 and 4 hours after taking the trial medication
  Painscore at rest (VAS)at time 1, 2, 3 and 4 hours, calculated as area under curve (AUC) from 1-4 hours after taking the trial medication.
Painscore during mobilization | 1, 2, 3 and 4 hours after taking the trial medication
  Painscore during active mobilization (VAS scale) defined by a standarized movement from recumbent position to sitting on the bedside at time 1, 2, 3 and 4 hours, calculated as area under curve (AUC) from 1-4 hours after taking the trial medication.
Degree of nausea | 1, 2, 3 and 4 hours after taking the trial medication
  Degree of nausea 1, 2, 3 and 4 hours after taking the trial medication.
Zofran consumption | 4 hours after taking the trial medication
  Consumption of Zofran (milligram) 0-4 hours after taking the trial medication.
Degree of dizziness | 1, 2, 3 and 4 hours after taking the trial medication
  Degree of dizziness 1, 2, 3 and 4 hours after taking the trial medication.
Incidence of vomiting | 0-4 hours after taking the trial medication
  Total number of vomits 0-4 hours after taking the trial medication.
Degree of sedation | 1, 2, 3 and 4 hours after taking the trial medication
  Degree of sedation 1, 2, 3 and 4 hours after taking the trial medication.

CONTACTS AND LOCATIONS:
Overall Officials: Rikke Soennichsen, MD, Principal Investigator — Glostrup University Hospital
Locations (1):
- Glostrup University Hospital, Glostrup Municipality, Glostrup, Denmark